CLINICAL TRIAL: NCT04410770
Title: Use of a Mood Tracker Smartphone App as a Chronic Health Management Intervention for Emotional Distress in Persons With TBI
Brief Title: Mood Tracker Smartphone App for Management of Emotional Distress After TBI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Memorial Hermann Health System (Other)
Collaborators: TIRR Memorial Hermann (Other); Baylor College of Medicine (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 90DPTB0016
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Emotional Distress
Keywords: Traumatic Brain Injury, Self-management, depression, anxiety, smart phone app
MeSH Terms: conditions — Brain Injuries, Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group, single masked, controlled trial with cross-over
Who Masked: Investigator, Outcomes Assessor
Masking Description: The clinical coordinator screens, consents, and completes baseline assessments with the participants. The clinical coordinator passes on the participants to the counselor who completes the support calls. The clinical coordinator and the counselor are unmasked. The participant is unmasked as he/she is aware of when he/she is receiving the support calls and when he/she is not. The 6 and 12 week outcomes are collected by a separate research assistant who is masked. The investigators are not exposed to the randomization process and are unaware of which arm the participant is assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (Active Comparator): Participants assigned to the active treatment arm are trained to use the mood tracker app and instructed to complete multiple self-ratings each week. Each the participant receives a support call each week for 6 weeks to engage the participant in the study and to address any problems the participant may have in completing self ratings. After 6 weeks of self-ratings, the participant complete the 6 week outcome. The participant is encouraged to continue completing the self-ratings, but does not receive any more support calls. After 6 more weeks, the 12 week outcome is assessed the participant's involvement with the study ends.
  Interventions: Behavioral: Mood tracker ratings
- Wait list (No Intervention): Wait list participants have no study activities for 6 weeks after completing the baseline assessment. After 6 weeks, list participants complete the 6 week assessment. After completing the assessment. wait list participants are trained to use the mood tracker app and instructed to complete multiple self-ratings each week. Each the participant receives a support call each week for 6 weeks to engage the participant in the study and to address any problems the participant may have in completing self ratings. After 6 weeks of self-ratings, the participant complete the 12 week outcome and the participant's involvement with the study ends.

INTERVENTIONS:
Behavioral: Mood tracker ratings — The participant rates his/her emotional distress several times a week using a specially developed smart phone app. The participant receives support call to ensure that self-ratings are being completed.
  Arms: Active intervention

SUMMARY:
Traumatic brain injury (TBI) is a common type of injury that affects thousands of people a year. TBI can cause a number of disabilities such as impaired cognition, decreased strength, decreased balance, problems controlling feelings, and difficulty communicating with others. Other problems that persons with TBI can have in the period after hospital discharge are anxiety and depress. These problems are common. At about one year after being injured, 44% of people have anxiety and 40% have depression. By five years after injury, 28% have depression and 17% have anxiety. If we think of emotional distress as having depression, anxiety, or both, at one year, 53% of people with TBI have emotional distress and, at five years, 38% have emotional distress. Many people with TBI are reluctant to seek help for emotional problems and when they do want help, it is hard to find. Many states have a shortage of mental health providers, many injured persons lack insurance that would pay for mental health treatment, and treatment may only be available a long distance from where people live.

In an attempt to address this problem, we are conducting a study designed to determine whether a self-management strategy can improve emotional distress or make emotional distress less like to develop. Previous studies have shown that simply keeping track of a problem may improve it. For example, tracking how often one has headaches can result in fewer headaches. Keeping track of one's blood pressure can lead to lower blood pressure. We are conducting this study to see if tracking one's level of emotional distress will result in lower levels of emotional distress. We are asking people with TBI to rate their levels of emotional distress several times a week using a special smart phone app. We will then conduct statistical tests to see if completing these ratings can cause people to have less emotional distress or prevent emotional distress from developing.

DETAILED DESCRIPTION:
Self-management Challenges for Persons with TBI:

A coordinated approach to chronic health management has been shown to be effective for a number of conditions such as asthma, (Wolf, et al., 2002) diabetes, (Glasgow, Funnell, et al., 2002) heart failure, (Glasgow, et al., 2002) and excess alcohol use (Hospital MM, Wagner, et al., 2016) among many others. Favorable results have been obtained across a wide range of clinical populations including adults (Glasgow et al., 2002) and children. (Hospital et al., 2016) The self-management aspect of chronic health management is often referred to as enablement. The patient is empowered to take action to improve his/her own health status. (Battersby, Von Korff, et al., 2010) Steps taken to facilitate this process are called self-management support. A wide range of self-management strategies have been used to improve health outcomes. These include skill-based training, goal setting, involvement with community based programs that provide education and support, self-monitoring, and use of technologies such as web-based content, text messages, graphic computer based feedback as opposed to verbal feedback, and others. (Battersby, Von Korff, et al., 2010) As reviewed in the Importance of the Problem section, persons with TBI have increased risk for a number of physical, cognitive, behavioral, and emotional co-morbidities that can decrease health and function, community living, and participation outcomes including employment. Given the limited availability and poor accessibility of psychiatric, psychological, counseling, and other mental health services, emotional distress is a particular concern for persons with TBI and their families. A number of studies have found that clinically significant emotional distress (defined here as depression, anxiety, or co-morbid depression and anxiety) is common after TBI. Depression and anxiety are more common in persons with TBI than in persons without TBI across all age ranges and all injury severities. (Osborn, Mathias, et al., 2016; Dikmen, Bombardier, et al., 2004) While anxiety may be more common early post-injury, depression is more problematic in the later years post-injury. (Always, Gould, et al., 2016) In this study, 40.1% of persons with TBI met diagnostic criteria for a depressive disorder at one year post-injury, while 44.1% had an anxiety disorder. By 5 years post-injury, 27.7% had depression and 16.8% had anxiety. If psychological distress is operationalized as anxiety, depression, or both, at year 1, 53.3% had psychological distress and at year 5, 33.7% had psychological distress. Anxiety and depression after TBI are associated with decreased social participation, limited independence in community living, decreased participation including employment, and low life satisfaction.

The frequent occurrence and negative impact of emotional distress after TBI is compounded by limited availability of mental health care providers and limited ability to access mental health services due to inability to pay and attitudinal barriers. Persons without TBI face challenges in obtaining mental health care. Findings from the National Comorbidity Survey Replication of 9,282 persons selected to represent the general population of the U.S. indicated that 1,350 (14.5%) met diagnostic criteria for a psychiatric disorder. Of these, 783 did not seek care for their psychiatric symptoms. (Mojtabi, Olfson, et al., 2011) Of those not seeking care, 44.8% did not perceive that they needed mental health services even though they met diagnostic criteria. The remaining 55.2% perceived that they needed care, but did not seek care due to various barriers. Structural barriers included inadequate financial resources, limited availability of providers, lack of transportation, and perceived inconvenience. Attitudinal barriers were experienced by about 4 times as many persons as structural barriers. Attitudinal barriers included perceived ineffectiveness of mental health services, stigma, and others. (Mojtabi, et al., 2011) These findings are of particular concern for our Center that serves the greater Houston metropolitan area, outlying areas in Texas, and various out of state and international constituencies. As reviewed in Section A - Importance of the Problem, Texas ranks in the lower 10% of all states in access to mental health care, persons needing mental health services who have insurance, and availability of mental health providers. (Mental Health in America, 2017) Poor accessibility of mental health services due to poor availability, cost of care, and various attitudinal barriers indicates the need for alternative service delivery models. Some encouragement is provided by a recent study (Bernecker, Banschback, et al., 2017) that found that of persons who needed mental health interventions but indicated that they would not use traditional psychotherapy even if they had an available provider and ability to pay, 51% indicated that they would be open to trying a web-based utility that would provide self-help and peer-support. Persons with TBI are even more challenged in accessing mental health services than the general population due to having more limited transportation options, being less likely to have healthcare coverage, and an even greater shortage of specialized providers.

Use of Technologic Solutions to Provide Mental Health Services in the Context of Health Management and Treatment of Emotional Distress in Persons with TBI:

The chronic health management literature provides a number of examples of electronic technologies used to support patient use of self-management strategies. In an intervention to decrease underage drinking, teens received text messages providing information about negative consequences of alcohol use, prompts to enhance self-efficacy, and social support. (Hospital et al., 2016) Teens receiving these messages showed greater interest in decreasing alcohol use than those who received control messages. A web based program was used to increase patient behavioral activation in an effort to increase self-management behaviors in a cohort including persons with asthma, hypertension, or diabetes. (Solomon, Wagner, Goes, 2012) Patients receiving this intervention showed greater increases in behavioral activation as indicated by higher self-efficacy and more regular tracking of health indicators such as medication compliance, glucose levels, and blood pressure than those not receiving the intervention.

In the psychotherapy literature, behavioral activation is often used as an intervention to decrease emotional distress. (Kanter, Manos, Bowe, et al., 2010) Key elements of behavioral activation include activity monitoring, assessment of life goals and values, activity scheduling, skills training, relaxation training, contingency management, procedures targeting verbal behavior, and procedures targeting avoidance. While these interventions are normally provided as a coordinated, comprehensive treatment, investigations have shown that self-monitoring of level of emotional distress is effective in improving mood. (Harmon, Nelson, Hayes, 1980; Manos, Kanter, Luo, 2011) In a different context, self-monitoring of risky behaviors in persons living with HIV has been shown to be an effective intervention to reduce these behaviors. (Lightfoot, Rotheram-Borus, et al., 2007) Given the high level of availability of smart phone technology throughout American society and the extensive familiarity with use of this technology possessed by most persons, smart phone based apps offer an attractive platform for providing low cost, easily assessed interventions for emotional distress in persons with TBI. Interventions provided through this medium are not be limited by barriers such as limited availability of providers, inability to afford care, perceived stigma of accessing care in office settings, and perceived inconvenience and ineffectiveness of standard office/clinic based mental services.

In a recent systematic review of smartphone apps used to address mental health issues, Donker and colleages (2013) determined that there are over 3,000 mental health related apps available for download. In aggregate, these apps have been downloaded hundreds of thousands of times. However, the systematic review revealed only 8 investigations of the effectiveness of these interventions. While findings were mixed, there was preliminary evidence that interventions delivered using this technology can cause clinically meaningful reductions in anxiety and depression. (Donker et al.,2013) Investigations of the use of these technologies to address emotional distress in persons with TBI are even more rare. Suffoletto and colleagues (2013) used educational text messages and symptom monitoring to reduce post-concussive symptoms in persons with mild TBI. Analyses revealed trends for reduction of severity for all symptoms over time but none of the effects was significant perhaps due to inadequate power. All participants believed the text messages were at least somewhat helpful. In another investigation, a smartphone app was used to monitor levels of depression and anxiety in 17 persons with TBI. (Juengst, Graham, et al., 2015) Self-ratings on the app were compared to results from assessments conducted by telephone. Among all 17 participants, 73.4% of scheduled app based assessments were completed indicating good compliance. Participants were generally satisfied with the experience of using the app. Self-ratings on the app were strongly correlated (0.81 to 0.91) with results of assessments conducted by phone. These findings indicate that this app has potential for use in ongoing monitoring, but the possible of effect of self-monitoring on severity of symptoms was not assessed.

Rationale for Proposed Study:

The current view of TBI as a chronic health condition indicates the need for long-term coordinated follow-up using principles of Chronic Care Management to identify late complications when they occur and provide appropriate interventions including self-management strategies. Emotional distress is a very common late complication that occurs with greater frequency for persons with TBI than for persons from the general population. Emotional distress in persons with TBI is associated with decreased function, limited independence with community living, decreased participation in community activities including employment, and deceased life satisfaction. However, treatment of emotional distress is complicated by reluctance of affected persons to seek care, limited availability of mental health care providers, inaccessibility of care due to inability to pay, perceived stigma of receiving mental health services, and perceived ineffectiveness and inconvenience of mental health care. Smartphone based apps offer an attractive option for addressing these issues. Apps are low cost; most mental health apps are available as free downloads. Their use is not limited by the inadequate availability of providers. Since the inconvenience of using an app is limited, the burden for attempting treatment and receiving no benefit is minimized. As a result, the numbers of persons who decline to access care due to perceived inconvenience and ineffectiveness may be decreased. The perceived stigma of seeking mental health services may also be decreased when these services are provided in a minimally intrusive manner by an app. A recent investigation found that over half of persons who indicated that they would not seek traditional psychotherapy were willing to use an app to address problem areas. (Bernecker, Banschback, et al., 2017) Apps have been shown to be an effective technology for tracking severity of emotional distress and there is evidence that monitoring of emotional distress is an efficacious treatment for decreasing distress.

Our proposed local research project will contribute to a coherent, sustained effort on application of chronic health management principles to long-term care for persons with TBI and add new knowledge to the current state of the art in this area of research. The specific aims, hypotheses, planned intervention, target population, and methodology for our proposed project were informed by our state of the art review of the relevant scientific literature on self-management strategies as applied to persons with TBI. The plan for statistical analysis and sample size calculations were developed by our team biostatistician. As we describe below, we have access to a much larger potential pool of participants than we will need to screen in order reach our sample size target. The research design was informed by our previous clinical trials including a telemedicine trial using counseling provided by phone calls. The target of this trial was informed by numerous focus groups with persons with TBI and families who have identified emotional distress as a key concern in the post-acute period after injury. We also obtained feedback from persons with injury regarding ease of use of the mood tracker app. Data collection procedures and selection of measures were informed by the scientific literature and our prior experience with these procedures and measures. This investigation is at the Intervention Efficacy Stage of Research. This will be an initial investigation of a smartphone based technology to reduce emotional distress in persons with TBI. The investigation will test the feasibility and practicality of this type of intervention in this population. Findings will have implications for how this type of intervention can be modified to be provided in the most effective manner.

Based on this review, we propose to conduct a randomized controlled trial of a smartphone app based self-monitoring intervention augmented by brief supportive telephone calls to decrease emotional distress in persons with TBI. This trial will be registered with ClinicalTrials.gov.

Specific Aims and Hypotheses:

Specific Aim 1: Determine the efficacy of self-monitoring of emotional distress using a smartphone app with accompanying by supportive telephone calls to decrease emotional distress in persons with TBI.

Hypothesis 1: Persons receiving the intervention will show a greater decrease in emotional distress at the post-treatment assessment (time 1) for the intervention group and the 2nd baseline assessment for the waitlist control group (time 1) as compared to the 1st baseline assessment (time 0).

Hypothesis 2: Both groups will show a reduction in emotional distress compared to their baseline levels of distress assessed prior to the intervention. For the intervention group, time 1 will be compared to time 0 and for the waitlist control group, time 2 will be compared to time 1.

Specific Aim 2: Determine factors that determine the magnitude of treatment effect.

Hypothesis 1: Greater engagement with the smartphone app as indicated by higher numbers of times the app was used to rate the degree of emotional distress and more days that ratings were completed during the intervention phase of the trial will be associated with greater decrease in emotional distress.

Specific Aim 3: Determine the persistence of the reduction of emotional distress once telephone counseling calls are discontinued.

Hypothesis 1: The initial reduction in emotional distress will diminish over time with a tendency for level of emotional distress to return to baseline.

Hypothesis 2: Maintenance of the initial reduction in the degree of emotional distress will be greater for participants who continue to use the smartphone app regularly.

ELIGIBILITY:
Inclusion Criteria:

* Medically documented complicated mild, moderate, or severe TBI
* Previous assent to be contacted regarding TBI related studies
* One year or greater post-injury
* Age 18 to 62 years at time of screening
* Adequately fluent in English to complete an interview and all study measures
* Living in a residential setting in the community
* Has capacity to give consent to medical research
* Access to a smartphone with capacity to download and run the T2 Mood Tracker app
* Acknowledges some degree of emotional distress

Exclusion Criteria:

* Has capacity to give consent to medical research
* Access to a smartphone with capacity to download and run the T2 Mood Tracker app
* Acknowledges some degree of emotional distress

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-09-29 (Estimated)

PRIMARY OUTCOMES:
Personal Health Questionnaire - 9 (PHQ-9) and Global Anxiety Disorder - 7 (GAD-7) scores combined. | 6 weeks from baseline.
  Scores for the PHQ-9 range from 0 to 27 with higher scores indicating greater depression. Scores for the GAD-7 range from 0 to 21 with higher scores indicating greater anxiety. These are measures of depression and anxiety that were developed for public health research. Scores from the 2 measures are combined to form an index of emotional distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Hermann Hospital-Texas Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon direct request to one of the investigators after all planned papers are published or after 5 years after completion of data collection which ever comes first.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of all planned papers or 5 years after all data have been collected.
Access Criteria: Direct request to one of the investigator by an investigator with a specific clinical question who has the capability to carry a successful new analysis of the study data.

REFERENCES:
- [Derived] Wisinger AM, Juengst SB, Sander AM, Broomfield RR, Vos L, Williams MW, Sherer M. Dimensions of participation as predictors of satisfaction with roles and abilities after traumatic brain injury. Rehabil Psychol. 2025 Jul 3. doi: 10.1037/rep0000627. Online ahead of print. PMID 40608439